CLINICAL TRIAL: NCT06653855
Title: The Effect of Cupping on Spasticity and Function of the Lower Extremity During Rehabilitation After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scott Getsoian (Industry)
Collaborators: Governors State University (Other)
Responsible Party: Sponsor-Investigator, Scott Getsoian, Physical Therapist, Ascension Health
Organization: Ascension Health (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIL20240041
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Stroke Gait Rehabilitation
Keywords: Cupping; Spasticity; stroke; rehabilitation
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The physical therapist providing the standard physical therapy treatment and the outcomes assessment will be masked to group allocation. However, the therapist administering the cupping and placebo cupping treatments will not be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cupping group (Active Comparator): This group (arm) will receive the dry static cupping intervention, along with the standard physical therapy treatment.
  Interventions: Other: Dry Static Cupping; Other: Standard physical therapy treatment
- Placebo cupping group (Sham Comparator): This group (arm) will receive a placebo-form of cupping (low, and non-therapeutic pressure amount in the cups), along with the standard physical therapy treatment.
  Interventions: Other: Placebo cupping; Other: Standard physical therapy treatment

INTERVENTIONS:
Other: Dry Static Cupping — A myofascial decompression cupping set with a precision pressure pump will be used to perform dry static cupping to the adductor and hamstring muscle groups of the affected limb, using a negative pressure of 300mmHg for eight minutes each.
  Arms: Cupping group
Other: Placebo cupping — The same protocol will be used as stated for the Dry static cupping intervention, with the only difference being that the cup will be pumped to 50mmHg instead of 300mmHg.
  Arms: Placebo cupping group
Other: Standard physical therapy treatment — Treatment will consist of typical physical therapy interventions performed for patients with spasticity of the lower extremity after stroke. These may include, but not be limited to:
  * Balance exercise
  * Therapeutic exercise
  * Neuromuscular/muscular coordination exercise
  * Manual (hands on) therapy
  * Gait training
  The treating physical therapist is left with the autonomy of the standard physical therapy treatment (within the above stated groups of interventions) because patients with the diagnosis of stroke do not all present with the same type or level of impairment. Furthermore co-morbidities (e.g., hypertension) and/or functional level (wheelchair bound vs. independent ambulator) may necessitate different treatment strategies. Therefore, while the general categories of treatment will remain the same across all study patients, it is expected that the treating physical therapist provides patient-specific interventions.

SUMMARY:
Physical therapists use dry static cupping for the treatment of many conditions, including spasticity for patients post-stroke. While research better describes the effects of dry static cupping for patients with orthopedic conditions, information is lacking on central conditions, such as stroke and resulting spasticity.

DETAILED DESCRIPTION:
Cupping is an ancient alternative medicine. A common form of cupping, called dry static cupping, involves creating negative pressure inside a therapeutic cup. The cup is then placed on the skin, creating a light suction effect. In Eastern Medicine, cupping has been used to treat a variety of diseases. More recently, in Western society, cupping has been used after injury, and among other effects, has been found to improve blood volume and tissue oxygenation to an area. These effects have originally been thought to be peripheral in nature, occurring at the cupping site, hence, why cupping has been used for treatment for conditions like carpal tunnel syndrome, spinal pain, knee osteoarthritis, and other musculoskeletal conditions.

However, a recent systematic review found cupping to be beneficial for rehabilitation after stroke. These conclusions raise the question of a possible mechanism for cupping to improve impairments related to the central nervous system, such as spasticity after stroke. However, many of the studies to date have serious methodological flaws that limit the direct causation of cupping to the reduction of spasticity. As well, the majority of studies only involve the upper extremity. No study has yet looked at the therapeutic effects of dry static cupping on lower extremity spasticity reduction after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80
* Acute stroke (within 6 months of stroke), with spasticity & hemiparesis of LE
* Referred by doctor for rehabilitation for a stroke-related condition
* Attending Ascension Rehabilitation of Joliet for rehabilitation
* Able to read or verbally understand English or Spanish

Exclusion Criteria:

* Absent sensation of the areas to be cupped
* Significant cognitive impairment
* Pregnancy
* Prescription anticoagulant medications
* Blood clotting disorder
* Uncontrolled hypertension
* Uncontrolled diabetes
* Open wounds within the cupping area
* Current DVT
* Hematoma over the cupping area
* Fracture over the cupping area
* Active cancer within the cupping area
* Current use of Baclofen
* Current use of Botox
* Current use of an anti-spasticity medication

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | At enrollment and then at 1, 2, and 3 months of treatment.
  The Modified Ashworth Scale measures spasticity on a 0-4 ordinal scale, with higher scores indicating greater spasticity. The grade is determined by passively moving a joint/muscle through a high velocity unidirectional quick stretch. For this study, spasticity will be assessed for the hip adductors and hamstrings of the affected side.
  Equipment:
  Mat Table
  Administration:
  Patient is positioned in supine on a mat table.
  For Hip Adduction: Physical therapist passively moves the affected lower extremity into hip abduction quickly keeping the knee in extension.
  For Hamstrings: Physical therapist passively moves the hip to 90 degrees of flexion and allows the knee to bend into knee flexion. Then, the therapist passively moves the affected knee into extension quickly.

SECONDARY OUTCOMES:
Six-Minute Walk Test (6MWT) | At enrollment and then at 1, 2, and 3 months of treatment.
  The Six-minute Walk Test is a measure of aerobic capacity and gait. It is measured in feet on a ratio scale.
  Administration:
  The patient is instructed to walk down an unobstructed path for six minutes, while the physical therapist walks behind them with a stopwatch and rolling tape measure to monitor the time and steps of the patient during the test. The distance (in feet) that the patient walked, after six minutes, is used as the score for the test.
  To note: blood pressure will be taken before and after the test.
Timed Up and Go (TUG) Test | At enrollment and then at 1, 2, and 3 months of treatment.
  The TUG assesses mobility, ability, and fall risk in older adults. It is measured in seconds, on a ratio scale.
  Equipment:
  * Chair with armrests
  * Stopwatch
  * Marker to designate 10' turn around point
  Administration:
  * The patient sits in the chair
  * On the command "ready and go" the patient gets up from the chair, walks 10 feet at a comfortable and safe pace, turns, walks back to the chair and sits down.
  * Timing begins at the instruction "go" and stops when the patient is seated
  * The patient must use the same assistive device for each assessment time, but is able to complete the test with multiple devices or no device.
  * The physical therapist will demonstrate the activity to the patient.
Berg Balance Scale (BBS) | At enrollment and then at 1, 2, and 3 months of treatment.
  The Berg Balance Scale is a 14-item test that measures static balance and fall risk in adults. Each item is scored on a 0-4 ordinal scale. At conclusion of the 14 items, the score is tallied.
  Equipment: Chair with arms, Chair without arms, Mat, Stopwatch, Yardstick, Slipper/sandal, 7 ¾" step, Blind fold, Tape.
  Items (14):
  1. sitting to standing
  2. standing unsupported
  3. sitting unsupported with feet on floor
  4. standing to sitting
  5. transfers
  6. standing unsupported with eyes closed
  7. standing unsupported with feet together
  8. reaching forward with outstretched arm
  9. pick up object from floor
  10. turn to look behind over each shoulder
  11. turning 360 degrees
  12. dynamic weight shifting while standing unsupported
  13. standing unsupported one foot in front
  14. standing on one leg

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Rehabilitation of Joliet, Joliet, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim M, Han C ho. The effectiveness and safety of cupping therapy for stroke survivors: A systematic review and meta-analysis of randomized controlled trials. J Korean Med. 2021;42(4):75-101. doi:10.13048/jkm.21039
- [Background] Choi TY, Ang L, Ku B, Jun JH, Lee MS. Evidence Map of Cupping Therapy. J Clin Med. 2021 Apr 17;10(8):1750. doi: 10.3390/jcm10081750. PMID 33920643
- [Background] Pontes NS, Barbosa GM, Almeida Silva HJ, Scattone Silva R, Souza CG, Lins CAA, de Souza MC. Effects of dry cupping on pain, function and quality of life in women with knee osteoarthritis: a protocol for a sham-controlled randomised trial. BMJ Open. 2020 Dec 24;10(12):e039857. doi: 10.1136/bmjopen-2020-039857. PMID 33361075
- [Background] Shen WC, Jan YK, Liau BY, Lin Q, Wang S, Tai CC, Lung CW. Effectiveness of self-management of dry and wet cupping therapy for low back pain: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Dec 23;101(51):e32325. doi: 10.1097/MD.0000000000032325. PMID 36595746
- [Background] Michalsen A, Bock S, Ludtke R, Rampp T, Baecker M, Bachmann J, Langhorst J, Musial F, Dobos GJ. Effects of traditional cupping therapy in patients with carpal tunnel syndrome: a randomized controlled trial. J Pain. 2009 Jun;10(6):601-8. doi: 10.1016/j.jpain.2008.12.013. Epub 2009 Apr 19. PMID 19380259
- [Background] Kim JI, Lee MS, Lee DH, Boddy K, Ernst E. Cupping for treating pain: a systematic review. Evid Based Complement Alternat Med. 2011;2011:467014. doi: 10.1093/ecam/nep035. Epub 2011 Jun 23. PMID 19423657
- [Background] Al-Bedah A, Aboushanab TS, Alqaed M, et al. Classification of Cupping Therapy: A Tool for Modernization and Standardization. J Complement Altern Med Res. 2016;1(1):1-10. doi:10.9734/JOCAMR/2016/27222
- [Background] Qureshi NA, Ali GI, Abushanab TS, El-Olemy AT, Alqaed MS, El-Subai IS, Al-Bedah AMN. History of cupping (Hijama): a narrative review of literature. J Integr Med. 2017 May;15(3):172-181. doi: 10.1016/S2095-4964(17)60339-X. PMID 28494847